CLINICAL TRIAL: NCT03895229
Title: The Effect of Morning Versus Evening Administration on The Pharmacokinetics and Pharmacodynamics of Empagliflozin
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ain Shams University (Other)
Collaborators: Drug Research Centre, Cairo, Egypt (Other)
Responsible Party: Principal Investigator, Mohamed Raslan, Principal investigator, Ain Shams University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: EMP-RES-BES-1018/0011
Record Dates: First submitted 2019-03-26; First posted 2019-03-29 (Actual); Last update posted 2019-04-02 (Actual); Status verified 2019-04

CONDITIONS: Diabetes Mellitus; Pharmacokinetics; Pharmacodynamics
Keywords: Diabetes; Empagliflozin; Circadian rythm
MeSH Terms: conditions — Diabetes Mellitus | interventions — empagliflozin; Tablets

STUDY DESIGN:
Intervention Model Description: A single group of 16 subjects will receive a single oral dose of Empagliflozin 10 MG Oral Tablet [Jardiance] at the morning(Period I) and the same group will receive the same dose of the same drug at the evening(Period II) after a seven days washout period
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental Arm (Experimental): Subjects will receive a single oral dose of Empagliflozin 10 MG Oral Tablet [Jardiance]
  Interventions: Drug: Empagliflozin 10 MG Oral Tablet [Jardiance]

INTERVENTIONS:
Drug: Empagliflozin 10 MG Oral Tablet [Jardiance] — Empagliflozin is a sodium-glucose co-transporter 2 inhibitor approved for treatment of type 2 diabetes mellitus
  Other Names: Jardiance (Boehringer Ingelheim and Eli Lilly)

SUMMARY:
An Open-label, One way, Two period Comparative study To Determine The effect of Morning Versus Evening administration of Empagliflozin 10mg on Its Pharmacokinetics And Pharmacodynamics in Healthy Adults

DETAILED DESCRIPTION:
Sixteen(16) healthy subjects will receive a single oral dose of Empagliflozin at the evening(Period I) and after a seven days washout period, the same 16 subjects will receive a single oral dose of Empagliflozin at the morning(Period II).

In both Periods(I and II), blood samples will be collected from each volunteer ethylene diamine tetra-acetic acid(KEDTA) containing tubes prior to drug administration then samples will be obtained at 0.33, 0.67, 1, 1.25, 1.5, 1.75, 2, 2.5, 3, 4, 6, 8, 10, 12, 24 and 48 hours(h) after drug administration.

These samples will be centrifuged and the plasma harvested and stored at -80°C until assay.

Urine samples will be collected over the first 24h after oral administration of the drug with sampling being at the following intervals: 0 to 4h, 4 to 8h, 8-12h, 12 to 24hr.

ELIGIBILITY:
Inclusion Criteria:

* Subject is at least 18-45 years at screening.
* Subject has a Body Mass Index of 18 to 35 kg/m2.
* Subject are non smokers or moderate smokers(not more than 5 cigarettes per day)
* Subject is willing to participate and give their final written consent prior to the commencement of the study procedures
* Subject is in good age-appropriate health condition as established by medical history, physical examination, and results of biochemistry, hematology and urine analysis testing within 4 weeks prior to study.
* Subject has a normal blood pressure and pulse rate, according to the reference normal ranges

Exclusion Criteria:

* Treatment with any known enzyme-inducing/inhibiting agents within 30 days prior to the start of the study and throughout the study.
* Subjects who have taken any medication two weeks preceding of the trial starting date.
* Documented history of sensitivity/idiosyncrasy to medicinal products or excipients.
* Any prior surgery of the gastrointestinal tract that may interfere with drug absorption.
* Gastrointestinal diseases.
* Renal diseases.
* Cardiovascular diseases specially transient ischemic attacks and cardiac dysrhythmia .
* Pancreatic disease including diabetes.
* Hepatic diseases as hepatic failure, cirrhosis, galactose intolerance, fructose intolerance, glycogen storage diseases
* Hematological disease or pulmonary disease
* Abnormal laboratory values.
* Subjects who have donated blood or who have been involved in a drug study within 6 weeks preceding the start of the study.
* Positive HIV test.
* History of or current abuse of drugs, alcohol or solvents.
* Endocrine disorders as Pheochromocytoma, Addison disease, glucagon deficiency, carcinomas, extra-hepatic tumors
* Autoimmune disorders as Graves disease
* (Central nervous system (CNS) disorders

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2018-10-19 (Actual); Study Completion 2018-10-26 (Actual)

PRIMARY OUTCOMES:
Maximum drug concentration in plasma (Cmax) | 0 up to 4 hours
  Maximum drug concentration in plasma measured in (ng/ml)
Area under the plasma concentration-time curve from time 0 to 48 hours(h) (AUC0→48h) | From first sampling interval up to 48 hours
  Area under the plasma concentration-time curve from time 0 to time(t) measured in(ng.h/ml)
Time to Maximum drug concentration in plasma (tmax) | 0 up to 4 hours
  Time corresponding to maximum drug concentration in plasma measured in Hours(h)

SECONDARY OUTCOMES:
Cumulative Urinary Glucose Excreted over the first 24 hours (Cumulative UGE) | From 0 up to 24 hours
  The Cumulative amount of Glucose excreted in Urine over the first 24 hours after drug administration measured in Milligrams (mg)
Half life( t½) of drug in plasma | Up to 48 hours
  Half life of drug measured in Hours(hr)

CONTACTS AND LOCATIONS:
Overall Officials: Rana M Ali, MD student, Principal Investigator — Ainshams University; Nagwa A Sabry, phD, Study Director — Ainshams University
Locations (1):
- Drug research centre, Cairo, Egypt

REFERENCES:
- [Derived] ElDash RM, Raslan MA, Shaheen SM, Sabri NA. The effect of morning versus evening administration of empagliflozin on its pharmacokinetics and pharmacodynamics characteristics in healthy adults: a two-way crossover, non-randomised trial. F1000Res. 2021 Apr 26;10:321. doi: 10.12688/f1000research.51114.1. eCollection 2021. PMID 34123370